CLINICAL TRIAL: NCT05815693
Title: Evaluate the Effectiveness for Long-term Consequences of COVID-19 of Mindfulness-based Stress Reduction (MBSR)
Brief Title: Cognitive-behavioral Therapy for Mental Disorder in COVID-19 Survivors
Acronym: LONGCOVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Socio Sanitaria Territoriale di Lecco (Other)
Responsible Party: Principal Investigator, Vincenzo Damico, Registered Nurse (RN), Doctor of Philosophy (PhD), Department of Anesthesia and Critical Care, Azienda Socio Sanitaria Territoriale di Lecco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASST LECCO, DEP. ICU
Record Dates: First submitted 2023-04-11; First posted 2023-04-18 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Post Acute COVID-19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Mindfulness-Based Stress Reduction; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (No Intervention): usual care for anxiety, depression, chronic pain and insomnia
- Group 2 (Experimental): mindfulness-based stress reduction (MBSR) for anxiety, depression, chronic pain and insomnia
  Interventions: Behavioral: mindfulness-based stress reduction (MBSR) and cognitive behavioral therapy (CBT)

INTERVENTIONS:
Behavioral: mindfulness-based stress reduction (MBSR) and cognitive behavioral therapy (CBT) — Patients with long-term consequences of COVID-19 (Chronic pain, anxiety, depression or insomnia) enrolled and randomly assigned to receive MBSR (n = 63), or usual care (n = 62). MBSR (training in mindfulness meditation and yoga) were delivered in 12 months with 2-hour groups each 2 months. Usual care included anything care participants received such as drug therapy.
  Arms: Group 2

SUMMARY:
The consequences of the Intensive Care Unit and the Covid-19 disease are still uncertain. However, many studies are bringing out often psychological and dramatic consequences for many COVID-survivor patients.

Among the ex-covid patients discharged from our Intensive Care Unit and with at least one covid-related psychological consequence, we want to evaluate the effectiveness for long-term consequences of COVID-19 of mindfulness-based stress reduction (MBSR) or usual care.

DETAILED DESCRIPTION:
Randomized controlled clinical study. All patients who survived COVID-19 and discharged from the intensive care unit of the Lecco hospital will be enrolled if present: chronic pain, anxiety, depression and/or insomnia in pharmacological therapy A group of patients will be observed during 12 months and evaluated with rating scales for chronic pain, anxiety, depression and insomnia.

The second (experimental) group will receive psychotherapy (mindfulness-based stress reduction and cognitive behavioral therapy) in addition to the pharmacological therapy

ELIGIBILITY:
Inclusion Criteria:

* Intensive care survivors
* Surviving COVID-19 patients
* Patients with Chronic Pain Anxiety Depression and/or Insomnia in drug therapy

Exclusion Criteria:

* Patients with Chronic Pain Anxiety Depression and/or Insomnia NOT in drug therapy
* Patients not hospitalized in intensive care for COVID-19

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Chronic pain | 6 months and 1 year
  pain that persists or recurs for longer than 3 months, and it exerts an enormous personal and economic burden, affecting more than 30% of people worldwide
Anxiety | 6 months and 1 year
  an emotion characterized by feelings of tension, worried thoughts, and physical changes like increased blood pressure
Depression | 6 months and 1 year
  a depressed mood or loss of pleasure or interest in activities for long periods of time
Insomnia | 6 months and 1 year
  a common sleep disorder that can make it hard to fall asleep, hard to stay asleep, or cause you to wake up too early and not be able to get back to sleep

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Damico, Principal Investigator — Azienda Socio Sanitaria Territoriale di Lecco
Locations (1):
- ASST Lecco, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No